CLINICAL TRIAL: NCT04703439
Title: A Mobile Phone Based Medication Reminder Program for Patients With Coronary Heart Diseases: A Pilot Study
Brief Title: An mHealth Intervention to Improve Medication Adherence and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00073395_1
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2021-01

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This group consisted of 116 participants who received a medication-taking reminder every morning at a random time between 7-8 am on WeChat app. Also, participants received a piece of educational material every five days at a random time between 8 am and 9 am regarding improving medication adherence and preventing coronary heart disease.
  Interventions: Behavioral: Medication-taking reminders & educational materials
- Control group (Placebo Comparator): This group consisted of 114 participants who only received a piece of educational material every five days at a random time between 8 am and 9 am. The educational materials sent to this group were general medical information, which were not specifically about improving medication adherence or preventing coronary heart disease.
  Interventions: Behavioral: Educational materials

INTERVENTIONS:
Behavioral: Medication-taking reminders & educational materials — The intervention has been described in arm/group descriptions, which lasted for 60 days for each participants.
  Arms: Experimental group
Behavioral: Educational materials — The intervention has been described in arm/group descriptions, which lasted for 60 days for each participants.
  Arms: Control group

SUMMARY:
Investigators evaluated the efficacy of a pilot-tested mHealth intervention to improving medication adherence and health outcomes among patients with coronary heart disease.

DETAILED DESCRIPTION:
This was a two-arm parallel randomized controlled trial, in which 116 and 114 participants were assigned to the experimental and control groups, respectively. The mHealth intervention in this study had been pilot tested and tailored. Specifically, the experimental group received a medication-taking reminder every morning via WeChat app and educational materials of coronary heart disease and medication adherence every five days via Message Express app. The control group received only general educational materials, which were irrelevant to coronary heart disease or medication adherence, every 5 days via Message Express app. All participants were diagnosed with coronary heart disease. The specific recruitment criteria of participants had been published in peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* (1) had a medical diagnosis of coronary heart disease;
* (2) aged 18 years or older;
* (3) had an antihypertensive medication regimen for 90 days or more from enrollment;
* (4) able to read messages through mobile phone;
* (5) had a mobile phone that could receive messages from WeChat and reminders from Message Express;
* (6) capable of giving his/her own consent; and
* (7) had an electronic blood pressure cuff to check blood pressures and heart rates.

Exclusion Criteria:

* was enrolled in other research studies

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change of medication non-adherence | Participants' medication non-adherence scores were measured at enrollment (baseline), 15-day, 30-day, 45-day, 60-day (end of intervention), 75-day, and 90-day (end of follow-up)
  Participants' medication non-adherence scores were measured using the Voils Medication Non-Adherence Extent Scale. Specifically, participants received the question items of the Voils Medication Non-Adherence Extent Scale every 15 days on WeChat app and provided answers
Change of systolic blood pressure | At enrollment (baseline), 15-day, 30-day, 45-day, 60-day (end of intervention), 75-day, and 90-day (end of follow-up)
  Participants self-measured their systolic blood pressures every 15 days using a blood pressure cuff and reported them to investigators
Change of diastolic blood pressure | At enrollment (baseline), 15-day, 30-day, 45-day, 60-day (end of intervention), 75-day, and 90-day (end of follow-up)
  Participants self-measured their diastolic blood pressures every 15 days using a blood pressure cuff and reported them to investigators
Change of heart rate | At enrollment (baseline), 15-day, 30-day, 45-day, 60-day (end of intervention), 75-day, and 90-day (end of follow-up)
  Participants self-measured their heart rates every 15 days using a blood pressure cuff and reported them to investigators

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Ryan Shaw, PhD, Study Chair — Duke University
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ni Z, Wu B, Yang Q, Yan LL, Liu C, Shaw RJ. An mHealth Intervention to Improve Medication Adherence and Health Outcomes Among Patients With Coronary Heart Disease: Randomized Controlled Trial. J Med Internet Res. 2022 Mar 9;24(3):e27202. doi: 10.2196/27202. PMID 35262490